CLINICAL TRIAL: NCT03207607
Title: The Effect of Mid-Morning Gel Snacks on Subjective Appetite, Glycemic and Insulin Responses, and Food Intake in Healthy Adults
Brief Title: Mid-morning Gel Snacks on Subjective Appetite, Glycemic and Insulin Responses, and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: The Hershey Company (Industry)
Responsible Party: Principal Investigator, Nick Bellissimo, PhD, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: REB2015-405
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Satiety; Food Intake
Keywords: Adults; Snacks; Appetite; Blood glucose; Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Coded snacks in shaded tetrapaks were provided to participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control snack (Experimental): Participants received control snacks prepared by real fruits (pear, orange and mango)
  Interventions: Other: Control snack
- Maltodextrin snack (Experimental): Participants received maltodextrin snacks (maltodextrin + control snack)
  Interventions: Other: Maltodextrin snack
- Whey protein snack (Experimental): Participants received whey protein snacks (whey protein + control snack)
  Interventions: Other: Whey protein snack
- Oat snack (Experimental): Participants received oat snacks (oat + maltodextrin + control snack)
  Interventions: Other: Oat snack
- Coconut oil snack (Experimental): Participants received coconut oil snacks (coconut oil + control snack)
  Interventions: Other: Coconut oil snack
- Snack skipping (Experimental): Participants received snack skipping
  Interventions: Other: Snack skipping

INTERVENTIONS:
Other: Control snack — Isovolumetric (238.4g) gel snack prepared by real fruits (186.2kcal)
  Arms: Control snack
Other: Maltodextrin snack — Isovolumetric (238.4g) gel snack with maltodextrin (271.8kcal)
  Arms: Maltodextrin snack
Other: Whey protein snack — Isovolumetric (238.4g) gel snack with whey protein (201.8kcal)
  Arms: Whey protein snack
Other: Oat snack — Isovolumetric (238.4g) gel snack with oats and maltodextrin (275.8kcal)
  Arms: Oat snack
Other: Coconut oil snack — Isovolumetric (238.4g) gel snack with coconut oil (276.4kcal)
  Arms: Coconut oil snack
Other: Snack skipping — no snack
  Arms: Snack skipping

SUMMARY:
The purpose of this study was to determine the effect of mid-morning gel snacks on subjective appetite, glucose and insulin responses, and food intake in healthy weight young adults.

DETAILED DESCRIPTION:
23 (14 male, 9 female) healthy, non-smoking human subjects aged 18-30 years with a body mass index (BMI) between 20 and 24.9 were recruited in the experiment. Five gel snacks including a control snack and four modified snacks containing whey protein, oats, coconut oil or maltodextrin were tested. On six separate mornings, at least 3 days apart and after a 12 hours overnight fast, each participant consumed a standardized breakfast of cereal, milk, and orange juice at home, then arrived in the lab 2 hours after breakfast to receive one of the five test snack treatments or skip snack. Subjective appetite by a 100 mm visual analogue scale (VAS) was measured at baseline (0 min) and after each treatment up to 2 h (15, 30, 60, 90, and 120 min). Blood glucose and insulin concentrations were measured via finger-prick at the same time VAS measurements were taken. Food intake was measured via ad libitum pizza lunch.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 30 years of age
* be healthy, non-smoking and not be taking any medications, including birth control
* body mass index (BMI) between 20 and 24.9

Exclusion Criteria:

* fasting plasma glucose >5.5 mmol/L
* health problems including previously diagnosed diabetes, known or uncertain pregnancy status at screening, gastrointestinal disease, liver or kidney disease
* major medical or surgical event within the past 6 months
* current or recent dieting
* breakfast skipping
* receiving any medications
* menstrual irregularities
* food sensitivities, allergies, intolerances, or dietary restrictions to foods including: cereal, orange juice, dairy, oat, coconut oil, honey, apple, pineapple, strawberry, and pear
* behavioural or emotional problems
* alcohol consumption >7 beverages/week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Subjective Appetite | Change from baseline over 120 minutes
  Participants completed subjective ratings on appetite (e.g., desire to eat, hunger, fullness, prospective food consumption) and well-being at baseline (0 min), 15, 30, 45, 60, 90, and 120 min after snack consumption, as well as immediately following lunch.

SECONDARY OUTCOMES:
Blood Glucose Response | Change from baseline over 120 minutes
  Blood was collected at baseline (0min), 15, 30, 45, 60, 90, and 120 min after snack consumption, as well as immediately following lunch to observe glycemic responses to gel snacks
Blood Insulin Response | Change from baseline over 120 minutes
  Blood was collected at baseline (0 min), 15, 30, 45, 60, 90, and 120 min after meal consumption, as well as immediately following lunch, to observe insulin responses to gel snacks
Food Intake | 30 min
  Participants consumed an ad libitum pizza lunch at 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University; Derick Rousseau, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada